CLINICAL TRIAL: NCT02239666
Title: A Prospective, Observational Study to Estimate the Proportion of Subjects With Plaque Psoriasis Who Achieve Complete Clearance on Biologics
Brief Title: Observational Study to Estimate the Effectiveness of Biologics When Treating Plaque Psoriasis
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: 20120363
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Plaque Psoriasis
Keywords: Dermatology, plaque psoriasis, biologic treatment, biologic naive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Moderate to Severe Plaque Psoriasis: Prospective cohort study of usual care for subjects initiating therapy for plaque psoriasis on approved biologic agents. A non-interventional study (NIS) of usual care over the 12 months following initiation of biologic therapy.
  Interventions: Other: NIS

INTERVENTIONS:
Other: NIS — This is a non-interventional study (NIS) of usual care over the 12 months following initiation of biologic therapy.

SUMMARY:
To estimate the real-world effectiveness of approved biologics in subjects with moderate-to-severe plaque psoriasis who are either starting or switching biologic medication.

DETAILED DESCRIPTION:
Plaque psoriasis is a chronic skin disease affecting 1-3% of US and European populations and severely impairs quality of life. Four biologics are authorized in Europe and the US for treatment of patients with moderate to severe psoriasis. Because complete skin clearance is rare with these agents, the treatment goal adopted by regulatory and reimbursement agencies is the proportion of patients achieving at least a 75% reduction from the subject's baseline PASI (Psoriasis Area and Severity Index) score or similarly, a sPGA [static Physician's Global Assessment) score of 0 or 1. Specifically, this study will provide information on the effectiveness of approved biologics as they are used in clinical practice. This information is currently not consistently available from other sources, including existing psoriasis patient registries.

Study Hypothesis: This study will estimate in each country the proportion of biologic treatment-naïve and biologic treatment-switching psoriasis subjects in the real-world having total clearance at 6 months after initiating a biologic.

The study population will include up to approximately 300 adults in each of up to 6 participating countries who have been diagnosed by their physicians with moderate to severe plaque psoriasis, and are initiating biologic therapy(biologic treatment-naïve or biologic treatment-switching) for plaque psoriasis.

Summary of Subject Eligibility Criteria: aged 18 or over; diagnosed with moderate to severe plaque psoriasis; initiating a biologic approved for psoriasis at study entry; able to fill out questionnaires; provided written informed consent; and not participating in a clinical trial utilizing an investigational agent in the 3 months prior to the first biologic dose.

Assessments: Skin clearance is the primary indicator of treatment effectiveness, and will be measured using the physician-reported PASI and sPGA. Other assessments will be by the following patient questionnaires: psoriasis symptom inventory (PSI), the dermatology life quality index (DLQI), the static patient's global assessment ( sPtGA), treatment satisfaction and global health status.

All subjects will be initiating biologic therapy at study entry. Therapy discontinuations, switches, and dosing changes during follow-up will be reported by the site and summarized.

Follow-up continues for approximately 12 months after first dose or until the subject is lost to follow-up or withdraws from the study (for any reason including death), whichever comes first. Where appropriate, data will be obtained for each subject during mandatory visits at 6 months (± 6 weeks) and 12 months (± 6 weeks) after first biologic dose, and at routine visits that occur during the follow-up period. To the extent possible data will also be collected at other usual care visits that occur during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* subjects who are greater than or equal to 18 YO diagnosed with moderate to severe plaque psoriasis
* subjects who will be initiating therapy with a biologic approved for moderate to severe psoriasis either for the first time (biologic treatment naive) or in course of switching to a different biologic agent
* subject who is able to complete questionnaires
* subject able to provide written informed consent

Exclusion Criteria:

- subjects who are participating in a clinical trial utilizing an investigational agent in the 3 months prior to the first biologic dose on study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults greater than or equal to 18 years of age who have been diagnosed with moderate to severe plaque psoriasis based on treating physician's judgment
Sampling Method: Non-Probability Sample
Enrollment: 899 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-01-05 (Actual)

PRIMARY OUTCOMES:
PASI100 | 6 months
  Physician-completed Psoriasis Area and Severity Index (PASI) measuring for each study subject average redness, thickness and scaliness of plaque psoriasis regions, weighted by area of involvement in each of four regions (head and neck, upper extremities, trunk, lower extremities). PASI100 represents a 100% improvement from baseline, that is, complete clearance. A static, or one-off, PASI (sPASI) score of 0 is equivalent to PASI100

SECONDARY OUTCOMES:
PASI100 (or sPASI=0) | 12 months
  Physician-completed Psoriasis Area and Severity Index (PASI) measuring for each study subject average redness, thickness and scaliness of plaque psoriasis regions, weighted by area of involvement in each of four regions (head and neck, upper extremities, trunk, lower extremities). PASI100 represents a 100% improvement from baseline, that is, complete clearance. A static, or one-off, PASI (sPASI) score of 0 is equivalent to PASI100
PASI100 (or sPASI=0) | 6 months and 12 months
  Physician-completed Psoriasis Area and Severity Index (PASI) measuring for each study subject average redness, thickness and scaliness of plaque psoriasis regions, weighted by area of involvement in each of four regions (head and neck, upper extremities, trunk, lower extremities). PASI100 represents a 100% improvement from baseline, that is, complete clearance. A static, or one-off, PASI (sPASI) score of 0 is equivalent to PASI100
sPGA=0 | 6 months and 12 months
  Physician-completed static Patient Global Assessment (sPGA) is a one-off assessment of severity of psoriasis on 6-point scale ranging from 0 (clear; no psoriasis) to 6 (very severe).
Psoriasis Symptom Inventory (PSI) responders | 6 months and 12 months
  A PSI responder is defined as a total PSI score less than or equal to 8, with no single item score more than 1
sPGA=0 or 1 | 6 months and 12 months
  Physician-completed static Patient Global Assessment (sPGA) is a one-off assessment of severity of psoriasis on 6-point scale ranging from 0 (clear; no psoriasis) to 6 (very severe).
PSI=0 | 6 months and 12 months
  Psoriasis Symptom Inventory (patient questionnaire) score of 0
Dermatology Life Quality Index (DLQI) =0 | 6 months and 12 months
  Measures functional disability of subjects with dermatological disorders. A self-administered 10-item questionnaire containing 6 functional scales (symptoms/feelings, sleep, leisure/daily activities, school/holidays, personal relationship and treatment).
Static Patient Global Assessment (sPtGA) | 6 months and 12 months
  Patient assessment of the severity of their psoriasis on a 6-point scale ranging from 0 (clear; no psoriasis) to 6 (very severe).
Percent PASI improvement (or sPASI scores) | 6 months and 12 months
  Physician-completed Psoriasis Area and Severity Index (PASI) measuring for each study subject average redness, thickness and scaliness of plaque psoriasis regions, weighted by area of involvement in each of four regions (head and neck, upper extremities, trunk, lower extremities). PASI score given represents a the percent improvement from baseline assessment. A static, or one-off, PASI (sPASI) score of 0 is equivalent to PASI100

CONTACTS AND LOCATIONS:
Overall Officials: Edward Hammond, Study Director — AstraZeneca
Locations (102):
- United States (37):
  - Research Site, Birmingham, Alabama
  - Research Site, Hot Springs, Arkansas
  - Research Site, Rogers, Arkansas
  - Research Site, Bakersfield, California
  - Research Site, Burbank, California
  - Research Site, Irvine, California
  - Research Site, Sacramento, California
  - Research Site, Aurora, Colorado
  - Research Site, Aventura, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Alpharetta, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Sandy Springs, Georgia
  - Research Site, Carmel, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Overland Park, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Owensboro, Kentucky
  - Research Site, Silver Spring, Maryland
  - Research Site, Clarkston, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, East Windsor, New Jersey
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Gahanna, Ohio
  - Research Site, Warren, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, West Jordan, Utah
  - Research Site, Norfolk, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Bridgeport, West Virginia
- France (17):
  - Research Site, Angers
  - Research Site, Argenteuil
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Chambray-lès-Tours
  - Research Site, Le Mans
  - Research Site, Limoges
  - Research Site, Lyon
  - Research Site, Nice
  - Research Site, Pierre-Bénite
  - Research Site, Poitiers
  - Research Site, Reims
  - Research Site, Rennes
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
- Germany (18):
  - Research Site, Bergen auf Rügen
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Buxtehude
  - Research Site, Dülmen
  - Research Site, Erlangen
  - Research Site, Eschweiler
  - Research Site, Friedrichshafen
  - Research Site, Gelsenkirchen-Feldmark
  - Research Site, Greifswald
  - Research Site, Hamburg
  - Research Site, München
  - Research Site, Münster
  - Research Site, Osnabrück
  - Research Site, Potsdam
  - Research Site, Quedlinburg
  - Research Site, Selters
  - Research Site, Simmern
- Italy (15):
  - Research Site, Ancona
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Cagliari
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Pavia
  - Research Site, Perugia
  - Research Site, Roma
  - Research Site, Roma (RM)
  - Research Site, Rome
  - Research Site, Siena
  - Research Site, Verona
- United Kingdom (15):
  - Research Site, Airdrie
  - Research Site, Cardiff
  - Research Site, Christchurch, Dorset
  - Research Site, Dundee
  - Research Site, Durham
  - Research Site, Exeter
  - Research Site, Lincoln
  - Research Site, London
  - Research Site, Nottingham
  - Research Site, Poole
  - Research Site, Portsmouth
  - Research Site, Redhill
  - Research Site, Scunthorpe
  - Research Site, Stourbridge
  - Research Site, Wolverhampton

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4136&filename=AZ_Brodalumab_Clinical_Study_Summary_Final.pdf